CLINICAL TRIAL: NCT03290105
Title: Efficacy of Chlorhexidine Mouth Wash in ICU Ventilated Patients: Microbiological Effects and Antiseptic Residual Concentrations
Brief Title: Microbial and Pharmacological Assessment of Chlorhexidine
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care, Hôpital Louis Mourier
Other Study IDs: HLM_JDR7
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Oropharynx Abnormality; Pneumonia, Ventilator-Associated; Chlorhexidine; Bacterium; Agent; Infection, Bacterial
Keywords: oropharyngeal colonization
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva for measurement of chlorhexidine concentration; swabbing of oropharyngeal secretions
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- study population: Consecutive critically-ill patients admitted to the ICU and receiving invasive mechanical ventilation for more than 48 hours

SUMMARY:
Ventilator-associated pneumonia (VAP) is the most frequent life-threatening nosocomial infection in the ICU. Oropharyngeal colonization with bacterial pathogens is the first step toward lung infection. Oral hygiene with Chlorhexidine mouth wash (CMW) is among the most widespread preventive measure to prevent VAP. Precise microbial documentation of CMW efficacy on oropharyngeal colonization is lacking. Investigators wish to determine CMW antimicrobial efficacy in ICU ventilated patients and to measure chlorhexidine residual concentration in patients' saliva at the same time-points after CMW.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is the most frequent life-threatening nosocomial infection in the ICU. Oropharyngeal colonization with bacterial pathogens is the first step toward lung infection. Oral hygiene with Chlorhexidine mouth wash (CMW) is among the most widespread preventive measure to prevent VAP. Although many guidelines and expert opinions recommend oral hygiene with chlorhexidine, optimal conditions of CMW use remain unknown. In addition, precise microbial documentation of CMW efficacy on oropharyngeal colonization is lacking. Investigators wish to determine CMW antimicrobial efficacy in ICU ventilated patients and to measure chlorhexidine residual concentration in the saliva at the same time-points after CMW.

In the participanting unit, CMW is performed every 6 hours with a 0.12% chlorhexidine solution.

Hence, microbial oropharyngeal sampling will be performed 6h after the last CMW (and just before the next one), to assess oropharyngeal colonization and then 15 minutes, 1 hour, 2 hours, 4 hours, and 6 hours after a new CMW to assess CMW efficacy in terms of bacterial growth.

In a subset of patients, 0.5 mL of saliva will be collected with a syringe at the same time points, with an additional T30 time (at 30 minutes) to measure chlorhexidine concentration.

ELIGIBILITY:
Inclusion Criteria:

* critically-ill patients admitted to the ICU and receiving invasive mechanical ventilation for more than 48 hours

Non-inclusion criteria:

* cervical or mouth surgery in the last 15 days;
* history of oropharyngeal neoplasm or of cervical or oropharyngeal radiotherapy,
* tracheotomy,
* age under 18

Exclusion Criteria:

* Patients whose samples retrieved less than 10 to the 3 colony forming unit (CFU)/mL bacteria and those who had two or more missing microbiological samples were secondarily excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Consecutive critically-ill patients admitted to the ICU and receiving invasive mechanical ventilation for more than 48 hours
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
changes over time of bacterial growth | 6 hours (360 minutes)
  oropharyngeal colonization (i.e., amount of bacterial growth in each oropharyngeal sample) before and after a mouth wash with chlorhexidine will be measured at different time points (before (H0) and 15 minutes, 60 minutes, 120 minutes, 240 minutes, and 360 minutes after the mouth wash with chlorhexidine)

SECONDARY OUTCOMES:
changes over time of bacterial growth of each bacterial specie | 6 hours (360 minutes)
  changes over time in bacterial growth of each bacterial species isolated in the oropharynx will be measured before (H0) and 15 minutes, 60 minutes, 120 minutes, 240 minutes, and 360 minutes after the mouth wash with chlorhexidine
susceptibility of isolates to chlorhexidine | 1 hour
  chlorhexidine minimal inhibitory concentration of dominant pathogens of each patient will be determined using the broth microdilution method recommended by the Clinical & Laboratory Standards Institute
salivary concentration of chlorhexidine | 6 hours (360 minutes)
  salivary concentration of chlorhexidine will be measured 15 minutes, 30 minutes, 60 minutes, 120 minutes, 240 minutes, and 360 minutes after the mouth wash with chlorhexidine using high-pressure liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Béatrice La Combe, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klompas M. Oropharyngeal Decontamination with Antiseptics to Prevent Ventilator-Associated Pneumonia: Rethinking the Benefits of Chlorhexidine. Semin Respir Crit Care Med. 2017 Jun;38(3):381-390. doi: 10.1055/s-0037-1602584. Epub 2017 Jun 4. PMID 28578560
- [Background] Klompas M, Speck K, Howell MD, Greene LR, Berenholtz SM. Reappraisal of routine oral care with chlorhexidine gluconate for patients receiving mechanical ventilation: systematic review and meta-analysis. JAMA Intern Med. 2014 May;174(5):751-61. doi: 10.1001/jamainternmed.2014.359. PMID 24663255